CLINICAL TRIAL: NCT05978427
Title: Efficacy and Safety of Superior Trunk Block Versus Interscalene Block for Post-operative Analgesia in Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: superior trunk vs interscalene
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2023-05

CONDITIONS: Superior Trunk Block Versus Interscalene Block for Post-operative Analgesia in Shoulder Surgeries
Keywords: superior trunk block; interscalene block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interscalene block group (Active Comparator): participants undergoing shoulder surgeries will receive ultrasound guided interscalene block
  Interventions: Procedure: interscalene block; Procedure: superior trunk block
- superior trunk block group (Active Comparator): participants undergoing shoulder surgeries will receive ultrasound guided superior trunk block
  Interventions: Procedure: interscalene block; Procedure: superior trunk block

INTERVENTIONS:
Procedure: interscalene block — will receive a 20 ml mixture of local anesthetic solution prepared as 10 ml of bupivacaine 0.5% diluted with 10 ml normal saline 0.9% will be injected in interscalene block.
Procedure: superior trunk block — will receive a 20 ml mixture of local anesthetic solution prepared as 10 ml of bupivacaine 0.5% diluted with 10 ml normal saline 0.9% will be injected in superior trunk block.

SUMMARY:
Efficacy and safety of superior trunk block versus interscalene block for post-operative analgesia in shoulder surgeries

DETAILED DESCRIPTION:
The interscalene brachial plexus block is the gold standard analgesic technique for surgery involving the shoulder and upper arm. However, due to its complications as hemidiaphragmatic paralysis, the superior trunk block was developed in an attempt to reduce major complications.The utility of the superior trunk block has yet to be studied in shoulder surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of Anaesthesiologists physical status (ASA) is I to II.
* Both genders.
* Aged group from 21 to 50 years old.
* Patients electively scheduled for shoulder surgery under general anesthesia with normal coagulation profile.

Exclusion Criteria:

* Refusal of the procedure or participation in the study.
* Any history or evidence of coagulopathy.
* Evidence of infection at injection site.
* Allergy to study drugs.
* Patients with pulmonary severe respiratory disease.
* Herniated cervical disc or cervical myelopathy.
* Pre-existing neuropathy of the operative limb

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
diaphragmatic paralysis postoperative | within 24 hours after surgery
  o The incidence of diaphragmatic paralysis postoperative assessed by Diaphragmatic excursion distance by Ultrasound

SECONDARY OUTCOMES:
analgesic efficacy | within 24 hours after surgery
  o Analgesic efficacy of the nerve block in both groups by assessing postoperative pain vas score
rescue analgesia | within 24 hours after surgery
  The total amount of rescue analgesia used
Post operative nausea and vomiting | within 24 hours after surgery
  incidence of post operative complications as nausea an vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided